CLINICAL TRIAL: NCT07024225
Title: Clinico-epidemiological and Endoscopic Characteristics of Patients With Colorectal Cancers : A Retrospective Study in Sohag, Egypt
Brief Title: Colorectal Cancers :A Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Khaled Abdelrahman Elsayed, Principal investigator, Sohag University
Other Study IDs: Soh-Med--25-5-8MS
Record Dates: First submitted 2025-05-28; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Clinical; Endoscopic; Pathological features
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with colorectal cancers: Patients more than 18 years old with colorectal cancers
  Interventions: Procedure: Endoscope

INTERVENTIONS:
Procedure: Endoscope — Lower endoscopy

SUMMARY:
Clinico-epidemiological and endoscopic characteristics of patients with colorectal cancers:A Retrospective study in Sohag

The aim :

1. determine the prevalence and clinicopathological pattern of patients with colorectal cancers
2. interpretative association between risk factors and severity of patient condition to define possible predictors
3. assess potential association between serum markers, imaging, endoscopic features and underlying condition.

DETAILED DESCRIPTION:
Methods :

1. all data will be obtained from patients as personal history (name, age, sex, occupation,residence , marital status, personal habits), history of illness at diagnosis, presence of diabetes or hypertension and other co-morbidity
2. general examination as general appearance,vital signs ,head and neck ,chest ,upper and lower limbs, Abdomen and pelvis ,and local examination as per rectal examination.
3. laboratory test as complete blood count and tumor markers ,imaging as abdominal ultrasound, CT,MRI, endoscopic findings and pathological features.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years old and above
* patients with confirmed diagnosis of colon or rectal cancer ,supported by histopathological result

Exclusion Criteria:

* patients with missed pathological or endoscopic data
* patients diagnosed with other malignancies rather than colorectal cancers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will be carried on patients more than 18 diagnosed as colon or rectal cancer supported by histopathological result
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of patients diagnosed with colon or rectal cancers within study period in sohag, Egypt | Retrospective review from 2015 to 2025
  To determine prevalence of colorectal cancers in sohag, Egypt
Correlation between baseline serum carcinoembryonic antigen (CEA) levels and tumor stage (TNM classification) | As recorded at diagnosis
  To assess the association between serum CEA levels and disease severity
Association between personal risk factors (e.g, age, sex, lifestyle habits, comorbidities) and tumor stage at diagnosis | based on initial diagnosis records from 2015 to 2025
  To identify risk factors associated with more advanced disease

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O Ahmed, Lecturer, Study Director — Sohag faculty of medicine, internal medicine department
Locations (1):
- Sohag faculty of medicine, Sohag, Sohag Government, Egypt

IPD SHARING:
Plan to Share IPD: No